CLINICAL TRIAL: NCT07088146
Title: Role of Intravenous Dexamethasone in Prolonging the Duration of Sub-Arachnoid Block in Pregnant Patients Undergoing Lower Segment Cesarean Section
Brief Title: Dexamethasone in Prolonging the Duration of Spinal Anesthesia Among Pregnant Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Huda Tariq, Principal Investigator, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201/IREF/RMU/2025
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Spinal Anesthesia; Post Operative Analgesia
Keywords: Adjuvants; Sub-Arachnoid Block; C-section
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone
- Group Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Immediately after sub-arachnoid block 8mg of Dexamethasone will be administered intravenously
  Arms: Group Dexamethasone
Drug: Placebo — 2ml of Normal saline will be given intravenously immediately after administration of spinal anesthesia
  Arms: Group Control

SUMMARY:
Lower segment C section is one of the most commonly performed surgeries worldwide. It is performed in spinal anesthesia. During Spinal Anesthesia a local anesthetic drug is administered in a space surrounding spinal cord and it blocks nerves originating from spinal cord providing both anesthesia and analgesia. This technique avoids harmful exposure of drugs to the baby inside the womb of mother. However this technique provides anesthesia and analgesia of limited duration which can be prolonged by addition of drugs to patient management regimen. One such drug is Dexamethasone which is a steroid commonly administered in the peri-operative period.

DETAILED DESCRIPTION:
To prolong the duration of Sub-Arachnoid block number of drugs which are known as adjuvants can be used. One of the commonly used adjuvant is Dexamethasone a steroid given by intravenous route having anti-emetic and anti-inflammatory effect. This drug also prolongs the duration of Sub-Arachnoid block which can be helpful in case of lengthy surgical procedure and also extends the duration of analgesia in the post operative period.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class: II and above.
* Elective Cesarean section under Spinal Anesthesia.

Exclusion Criteria:

* Gestational diabetes
* Body mass index >35 kg/m2
* Diabetes mellitus
* Adrenal insufficiency
* Chronically receiving steroids
* Allergic to study medications
* Sensory block level less than T4

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Time for block to regress by two dermatomes in post operative period | This will be the time in minutes from end of C section in post operative period for the block to regress by two dermatomes

SECONDARY OUTCOMES:
Time to rescue analgesia | This will be the time in minutes from the end of Cesarean section in the post operative period to first rescue analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Abeera Zareen, MBBS,FCPS, Study Chair — Rawalpindi Medical College
Locations (1):
- Benazir Bhutto Hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Wahab AH, Abd Alla ES, Abd El-Azeem T. Effect of intravenous dexamethasone on the duration of hyperbaric bupivacaine spinal anesthesia in lower abdominal surgery, Randomized controlled trial. BMC Anesthesiol. 2023 Sep 22;23(1):323. doi: 10.1186/s12871-023-02282-y. PMID 37736711
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10515039/